CLINICAL TRIAL: NCT00757991
Title: A Population Based Control Collection for Genetic Studies in East Anglia
Brief Title: Blood Samples From Healthy Volunteers for Genetic Studies in the East Anglia Region of the United Kingdom
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cancer Research UK (Other)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: CDR0000598880; MREC-SEARCH-CONTROL; MREC-07/MRE05/17
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2008-09

CONDITIONS: Healthy, no Evidence of Disease
Keywords: healthy, no evidence of disease
MeSH Terms: interventions — Amplified Fragment Length Polymorphism Analysis

INTERVENTIONS:
Genetic: polymorphism analysis
Other: laboratory biomarker analysis
Other: questionnaire administration

SUMMARY:
RATIONALE: Studying samples of blood from healthy volunteers in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This study is looking at genetic susceptibility to cancer and interactions between genes and the environment in healthy volunteers.

DETAILED DESCRIPTION:
OBJECTIVES:

* To obtain blood samples and simple epidemiological information on a population-based series of adult individuals without cancer.
* To establish whether polymorphisms in putative cancer predisposition genes are associated with an increased risk of cancer by comparing the frequency of alterations in these genes with the corresponding frequency in a comparable series of cancer patients.
* To examine the interactions between genetic and non-genetic risk factors.

OUTLINE: This is a multicenter study.

Participants complete a simple epidemiological questionnaire.

Participants undergo blood sample collection. DNA is extracted from these samples for polymorphism analysis of low penetrance cancer susceptibility genes in the following related clinical trials: MREC-SEARCH-CANCER, MREC-SEARCH-PROSTATE, and MREC-SEARCH-BREAST. They may also be used in the analyses of the following related clinical trials: MREC-SEARCH-OVARIAN, MREC-SEARCH-ENDOMETRIAL, MREC-SEARCH-COLORECTAL.

PROJECTED ACCRUAL: A total of 2,000 male and 2,000 female participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cancer-free participants randomly selected from the age-sex registry of a general practice in the East Anglia region of the United Kingdom

  * Two general practices from each district within East Anglia participate (up to 10 total participating practices)

PATIENT CHARACTERISTICS:

* Identified by the participant's general practitioner as fit to contact for this study
* No prior diagnosis of cancer
* No serious mental illness or retardation

PRIOR CONCURRENT THERAPY:

* Not specified

Ages: 35 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2008-02

PRIMARY OUTCOMES:
Acquisition of blood samples and epidemiological information
Investigation of whether polymorphisms in putative cancer predisposition genes are associated with an increased risk of cancer
Examination of the interactions between genetic and nongenetic risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Paul Pharoah, MD, Study Chair — Cancer Research UK
Locations (1):
- University of Cambridge Cancer Research UK, Cambridge, England, United Kingdom